CLINICAL TRIAL: NCT02578693
Title: Long Term Follow-up for Subjects With Chronic Hepatitis C Infection Who Received Interferon-based Therapy or Direct-acting Antiviral Agents (DAAs)-Based Therapy
Brief Title: Follow up of IFN Vs DAAs HCV SVR (IFDACS Study)
Status: Completed | Type: Observational
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: Beijing 302 Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Yamanashi Prefectural Central Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: H&H_HCV IFN Vs DAAs Fu
Record Dates: First submitted 2015-10-16; First posted 2015-10-19 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis C Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum/Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is designed to provide long term clinical and virologic follow up in subjects infected with hepatitis C virus (HCV) who received interferon-based therapy or direct-acting antiviral agents (DAAs)-based therapy. This long term follow up study is observational and no treatment is provided for HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C treated with interferon-based therapy or direct-acting agents (DAAs)-based regimen;
* Provide written, informed consent;
* Be willing and able to comply with the visit schedule and protocol-mandated procedures.

Exclusion Criteria:

* Individuals planning to start a new course of hepatitis C therapy including any investigational drug or device during the course of the follow-up time frame;
* History of clinically significant illness or any other major medical disorder that may interfere with follow up, assessments, or compliance with the protocol.
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects infected with hepatitis C virus (HCV) who received interferon-based therapy or direct-acting antiviral agents (DAAs)-based therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1210 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 36 months
  The primary outcome measure is the occurence (yes or no) of sustained virologic response (SVR), defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) in serum at least 3 months after stopping therapy. Point estimates and confidence intervals will be calculated to describe the frequency of SVR in various patients receiving IFN or DAAs based treatment.

SECONDARY OUTCOMES:
Treatment persistence | 36 months
  Treatment persistence will be the duration of treatment measured from the first dose of medication until treatment is discontinued. Reasons for premature discontinuation of treatment will be recorded.
Virological breakthrough | 36 months
  The occurrence of virological breakthrough defined as an increase of HCV RNA by at least 1-log over nadir or to >100 IU if previously undetectable.
Liver disease progression | Post treatment 10 years
  Liver disease progression is a composite endpoint measured by laboratory parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, albumin, platelets, prothrombin time (PT) and α-fetoprotein) and observed or reported clinical signs and symptoms.
Proportion of participants who develop hepatocellular carcinoma (HCC) through Year 10 by treatment regimen | Post treatment 5 years

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Humanity & Health Medical Centre
Locations (3):
- China (2):
  - Liver Fibrosis Diagnosis and Treatment Centre, 302 Hospital, Beijing, Beijing Municipality
  - Humanity and Health GI and Liver Centre, Hong Kong, Hong Kong
- Yamanashi Prefectural Central Hospital, Kofu, Yamanashi, Japan